CLINICAL TRIAL: NCT04907474
Title: A Study Evaluating Pupil Dilation Speed With the Micro-Array Print (MAP) Dispenser Comparing 2 Dosing Regimens of Tropicamide-Phenylephrine Fixed Combination Ophthalmic Solution
Brief Title: Evaluation of Pupil Dilation Speed With the MAP Dispenser
Acronym: SPEED
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Eyenovia Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Diagnostic
Other Study IDs: EYN-MYD-TP-41
Record Dates: First submitted 2021-05-25; First posted 2021-05-28 (Actual); Results first posted 2025-01-09 (Actual); Last update posted 2025-01-09 (Actual); Status verified 2025-01

CONDITIONS: Mydriasis
MeSH Terms: conditions — Mydriasis

STUDY DESIGN:
Intervention Model Description: All subjects received both treatments. Subjects were randomized to treatment order
Who Masked: Participant, Outcomes Assessor
Masking Description: Only 1 mist or 2 mists of the drug will be administered per treatment visit and will occur in a randomized sequence order using on of the two sequences AB or BA where A is 1 mist of the fixed combination and B is 2 mists of the fixed combination
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sequence AB (Other): Sequence AB: 1 mist of tropicamide-phenylephrine fixed combination solution administered to each eye with the Micro Array Print (MAP) Dispenser followed by 2 mists of tropicamide-phenylephrine fixed combination solution administered to each eye with the MAP Dispenser
  Interventions: Drug: tropicamide-phenylephrine fixed combination ophthalmic solution
- Sequence BA (Other): Sequence BA: 2 mists of tropicamide-phenylephrine fixed combination solution administered to each eye with the Micro Array Print (MAP) Dispenser followed by 1 mist of tropicamide-phenylephrine fixed combination solution administered to each eye with the MAP Dispenser
  Interventions: Drug: tropicamide-phenylephrine fixed combination ophthalmic solution

INTERVENTIONS:
Drug: tropicamide-phenylephrine fixed combination ophthalmic solution — Tropicamide-phenylephrine fixed combination ophthalmic solution is a tropical drug solution for mydriasis

SUMMARY:
1 mist or 2 mists of the study drug will be administered to both eyes according to a pre-specified randomization plan to determine the effect on pupil dilation

DETAILED DESCRIPTION:
After screening, eligible subjects will be scheduled for 2 treatment visits where either 1 mist or 2 mists of the study drug will be administered to both eyes according to a pre-specified randomization plan. Safety evaluations and efficacy measurements will be performed at specified time intervals thereafter.

Pupil dilation for each treatment will be compared at each time interval.

ELIGIBILITY:
Inclusion Criteria:

1. Photopic screening pupil diameter ≤ 3.5 mm in each eye

Exclusion Criteria:

1. Allergy to phenylephrine hydrochloride, tropicamide, or benzalkonium chloride.
2. Use of benzodiazepines, monoamine oxidase inhibitors, tricyclic antidepressants, anticonvulsants, cholinergic drug at screening or anticipated during the study period.
3. History of closed-angle glaucoma.
4. Anatomically narrow anterior chamber angles (Van Herrick grade ≤ 2 in either eye).
5. Ocular surgery or laser treatment of any kind prior to the Screening Visit.
6. History of iris trauma, surgery, or atrophy.
7. Irregularly-shaped pupil secondary to ocular trauma or congenital defect, or history of neurogenic pupil disorder.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2021-05-24 (Actual); Primary Completion 2021-06-03 (Actual); Study Completion 2021-06-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tsontcho Ianchulev, MD, MPH, Study Director — Eyenovia Inc.
Locations (1):
- CODET Vision Institute, Tijuana, Estado de Baja California, Mexico

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chayet A, Ramirez A, Scott B, Whitcomb J, Lam P, Ianchulev T. Pupil dilation evaluation of two mydriatic dosing profiles delivered by the Optejet(R). Ther Deliv. 2023 Feb;14(2):93-103. doi: 10.4155/tde-2022-0061. Epub 2023 May 9. PMID 37158245

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 61 subjects were consented at a single-center and assessed for eligibility. A total of 60 subjects met eligibility criteria and were randomized. (1 consented subject was ineligible). All eligible subjects received both treatments.A total of 60 subjects completed the study. No subjects were lost to follow-up or were terminated early from the study.
Groups:
- 1 Mist Then 2 Mists: 1 mist of tropicamide-phenylephrine fixed combination solution administered to each eye with the Micro Array Print (MAP) Dispenser followed by 2 mists of tropicamide-phenylephrine fixed combination solution administered to each eye with the Micro Array Print (MAP) Dispenser
- 2 Mists Then 1 Mist: 2 mists of tropicamide-phenylephrine fixed combination solution administered to each eye with the Micro Array Print (MAP) Dispenser followed by 1 mist of tropicamide-phenylephrine fixed combination solution administered to each eye with the Micro Array Print (MAP) Dispenser
Period: Overall Study
Arm/Group | 1 Mist Then 2 Mists | 2 Mists Then 1 Mist
Started | 31 | 30
Completed | 30 | 30
Not Completed | 1 | 0
Not completed — Not eligible for study per Inc/Exc and was not treated. Not included in analysis. | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Participants: Participants were administered either 1 Mist/Eye or 2 Mists/Eye of the study drug on separate days in the clinic occurring at least 4 days, but no more than 7 days apart.
Arm/Group | All Participants
Number analyzed (Participants) | 60
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.3 (14.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 37
  Male | 23
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 59
  Not Hispanic or Latino | 1
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 60
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  Mexico | 60

OUTCOME MEASURES:

1. Primary Outcome: Mean Change in Pupil Diameter From Baseline
Description: The primary performance endpoint is Mean Change in pupil diameter at 35 minutes versus per-visit baseline, as measured by digital pupillometry in highly photopic conditions. The highly photopic condition was established using a fully-charged transilluminator (muscle light) at the brightest setting.
Time Frame: 35 minutes post drug administration
Measure: Mean (Standard Deviation); unit: millimeters
Units Other Than Participants: Eyes
Groups:
- 1 Mist: One mist of tropicamide-phenylephrine fixed combination solution administered to each eye with the MAP Dispenser
  tropicamide-phenylephrine fixed combination ophthalmic solution: Tropicamide-phenylephrine fixed combination ophthalmic solution is a topical drug solution for mydriasis
- 2 Mists: Two mists of tropicamide-phenylephrine fixed combination solution administered to each eye with the MAP Dispenser
  tropicamide-phenylephrine fixed combination ophthalmic solution: Tropicamide-phenylephrine fixed combination ophthalmic solution is a topical drug solution for mydriasis
Arm/Group | 1 Mist | 2 Mists
Number analyzed (Participants) | 60 | 60
Number analyzed (Eyes) | 120 | 120
millimeters | 4.55 (.68) | 4.88 (.60)

ADVERSE EVENTS:
Time Frame: 7 days
Groups:
- 1 Mist Then 2 Mists: 1 mist of tropicamide-phenylephrine fixed combination solution administered to each eye with the MAP Dispenser followed by 2 mists of tropicamide-phenylephrine fixed combination solution administered to each eye with the MAP Dispenser
- 2 Mists Then 1 Mist: 2 mists of tropicamide-phenylephrine fixed combination solution administered to each eye with the MAP Dispenser followed by 1 mist of tropicamide-phenylephrine fixed combination solution administered to each eye with the MAP Dispenser
Arm/Group | 1 Mist Then 2 Mists | 2 Mists Then 1 Mist
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/30
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/30
Other Adverse Events (participants affected / at risk) | 0/30 | 0/30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-05-06): https://cdn.clinicaltrials.gov/large-docs/74/NCT04907474/Prot_SAP_000.pdf